CLINICAL TRIAL: NCT03932760
Title: Randomized Trial of Telehealth Group Intervention to Reduce Perinatal Depressive Symptoms in Diverse Populations
Brief Title: Telehealth Group Intervention for Perinatal Depressive Symptoms
Acronym: TePOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Gwen Latendresse, Assitant Dean, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00113917; R01NR017620 (NIH)
Record Dates: First submitted 2019-04-16; First posted 2019-05-01 (Actual); Results first posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Perinatal Depression

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UPLIFT Program (Experimental): Weekly one-hour group sessions for 10 weeks facilitated by a mental health professional.
  Interventions: Behavioral: UPLIFT Program
- Pregnancy Skills Group (Active Comparator): Weekly one-hour group sessions for 10 weeks facilitated by a registered nurse.
  Interventions: Behavioral: Attention Control Group

INTERVENTIONS:
Behavioral: UPLIFT Program — UPLIFT is based on cognitive behavioral therapy and mindfulness-based practices. Participants meet by videoconference using any electronic device (laptop, tablet, smart phone) from their own home.
  Arms: UPLIFT Program
Behavioral: Attention Control Group — Program is based on standard prenatal, childbirth, infant feeding, and parenting education curriculum. Participants meet by videoconference using any electronic device (laptop, tablet, smart phone) from their own home.
  Arms: Pregnancy Skills Group

SUMMARY:
The goal of the project is to evaluate for the first time, the effectiveness of using a telehealth approach to reducing perinatal depressive symptoms in diverse groups of childbearing women; urban and rural-dwelling, and from Hispanic and predominantly North European Descent populations. Pregnant women connect for one hour weekly, for 8 weeks, using their own electronic device, from whatever location they choose (e.g. home), to attend videoconference groups facilitated by a mental health professional. The approach is cost effective and reduces barriers to access to mental health services, particularly for women living in rural, low-resource, and minority communities, and those without adequate transportation, financial resources, childcare, or work release time.

DETAILED DESCRIPTION:
Perinatal depression (PD) affects 12-15% of women and contributes to adverse outcomes, e.g. preterm birth, low birth weight, and impaired cognitive development of the child. Screening optimizes the detection of PD, but does not reduce barriers to mental health services (MHS) encountered by women who screen positive. A known shortage of MHS across the nation is a significant barrier, particularly in low resource and rural settings. Telehealth is a promising approach to reducing barriers, but there is little research on the effectiveness of telehealth to reduce perinatal depressive symptoms (PDS). There is high potential for telehealth to deliver effective, lower cost MHS to childbearing women, particularly those in low resource settings.

The proposed project is a randomized controlled trial among women with mild to moderate PDS. The project aims to evaluate; 1) the effectiveness of a group mental health videoconference intervention (VCI) to reduce PDS across pregnancy and postpartum, and (2) differences in PDS between diverse groups of childbearing women: rural and urban-dwelling, and Latina and predominantly North European Descent (NED) populations. The investigators hypothesize that women participating in the VCI will have significantly lower PDS across pregnancy and postpartum than women in an equivalent attention control (AC) group, and the results will differ between diverse groups. A total of 192 women will be enrolled; 48 in each study group. Participants are randomly assigned to study groups: VCI +standard of care, or AC + standard of care. Sessions are delivered via Utah Telehealth Network (UTN). Women in both groups attend weekly one-hour group sessions for 8 weeks using any electronic device (laptop, tablet, smart phone) from their own home. PDS is measured six times throughout enrollment--Time 1 = pre-intervention; T2 = immediately following week 9 of group intervention classes (post-intervention), T3= 2 months post-intervention; T4= 4 months post-intervention; T5 = 6 months post-intervention; T6 = 8 post-intervention.

This study is the first to use a VCI to engage women in a facilitated group approach to reducing PDS, and to evaluate the impact among diverse groups. The approach is cost effective and reduces barriers to access to MHS, particularly for women living in low-resource, and minority communities, and those without adequate transportation, childcare, or work release time. The VCI can be replicated in any setting (e.g. rural or urban), and can be adapted to the needs of diverse communities. The study advances the field by establishing whether a group telehealth intervention reduces PDS, and whether this differs based on the population. If effective and implemented broadly, far fewer women and families would suffer the negative consequences of depression. The project is in line with NINR's high priority areas, including the use of technology to promote health, and a focus on self-management and symptom science.

ELIGIBILITY:
Inclusion Criteria:

* women age 18 and older
* have a viable pregnancy (any gestational age) or postpartum (up to 6 months)
* have an Edinburgh Postpartum Depression Scale (EPDS) score between 9 and 20
* are English or Spanish speaking
* are receiving clinical services at a collaborating prenatal or public health clinic associated with the U of Utah or Utah rural Health Districts

Exclusion Criteria:

* women who have an EPDS score less than 9 or greater than 20
* have a current diagnosis of a serious mental illness, such as psychosis, schizophrenia, bipolar disorder, severe depression, suicidal ideation, homicidal ideation
* begun taking or changed dosage of any medications for a mental health condition within the previous 6 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant and postpartum women
Enrollment: 99 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gwen Latendresse, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI will share de-identified data to other investigators for study, including demographics, outcomes, communication methodology, and design. Data will be shared with investigators working under an institution with a Federal Wide Assurance (FWA) and can be used for secondary study purposes. The PI agrees to make available data within one year of the completion of the funded project period and manuscripts pertaining to the aims. The PI agrees to share data in a manner that is fully consistent with NIH data sharing policies and applicable laws and regulations.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The PI agrees to make available data within one year of the completion of the funded project period
Access Criteria: Data will be shared with investigators working under an institution with a Federal Wide Assurance (FWA) and can be used for secondary study purposes.

REFERENCES:
- [Derived] Iacob E, Kausler R, Williams M, Simonsen S, Smid M, Weissinger K, Latendresse G. Protocol for a randomized controlled trial to evaluate the effectiveness of a telehealth group intervention to reduce perinatal depressive symptoms. Contemp Clin Trials. 2024 Dec;147:107738. doi: 10.1016/j.cct.2024.107738. Epub 2024 Nov 13. PMID 39542133

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the period from May 1, 2020 through May 31, 2022, 535 women were reached out to for participation in the study. Participants were recruited from University of Utah UHealth clinics as well as rural health districts.
Pre-assignment Details: Out of the 535 women reached out to, 331 were unable to be contacted after four attempts. Of the remaining 204, 58 were ineligible for a combination of non-mutually exclusive factors including mental health diagnoses (n= 35), medication changes in the last 6 weeks (n=15), >6 months postpartum (n=9), and other (n=6). Of the 147 who remained eligible to participate, 99 were consented. Of these, 17 were lost to contact prior to randomization, and 81participants were randomized.
Period: Overall Study
Arm/Group | UPLIFT Program | Pregnancy Skills Group
Started | 40 | 41
Baseline (Number of participants who completed survey at baseline.) | 36 | 33
Post (Number of participants who completed survey post intervention.) | 29 | 30
2 Months (Number of participants who completed survey at 2 months.) | 31 | 29
4 Months (Number of participants who completed survey at 4 months.) | 31 | 29
6 Months (Number of participants who completed survey at 6 months.) | 30 | 28
8 Months (Number of participants who completed survey at 8 months.) | 30 | 28
Completed | 32 | 30
Not Completed | 8 | 11
Not completed — Became Ineligible | 2 | 5
Not completed — Withdrawal by Subject | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UPLIFT Program | Pregnancy Skills Group | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 41 | 81
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 30 [19 to 41] | 31 [21 to 39] | 31 [19 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 41 | 81
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 8
  Not Hispanic or Latino | 28 | 28 | 56
  Unknown or Not Reported | 10 | 7 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 0 | 1
  White | 28 | 24 | 52
  More than one race | 3 | 5 | 8
  Unknown or Not Reported | 6 | 9 | 15
Region of Enrollment [Number; unit: participants]
  United States | 40 | 41 | 81

OUTCOME MEASURES:

1. Primary Outcome: Change in Depressive Symptoms Over Time
Description: Self-completed: Edinburgh Postnatal Depression Scale measures depression symptoms during pregnancy and postpartum. The instrument will measure depressive symptoms at 6 time points during pregnancy and postpartum. The instrument is on a scale of 0-30, with 0 indicating no symptoms, and 30 indicating the highest severity of symptoms. Scores < 10 = no depressive symptoms; 10-15 = mild; 16-20 = moderate; > 20 = severe.
Time Frame: Time 1 = pre-intervention (Baseline); T2 = immediately following week 9 of group intervention classes (Post), T3= 2 months post-intervention; T4= 4 months post-intervention; T5 = 6 months post-intervention; T6 = 8 post-intervention
Population: Number Analyzed differs from Overall Number of Participants Analyzed due to participants becoming ineligible, withdrawing, and opting to not complete surveys at certain time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | UPLIFT Program | Pregnancy Skills Group
Number analyzed (Participants) | 40 | 41
units on a scale
  Baseline: number analyzed (Participants) | 36 | 33
  Baseline | 11.11 (3.85) | 10.52 (4.52)
  Post: number analyzed (Participants) | 29 | 30
  Post | 7.34 (2.79) | 7.69 (3.92)
  2 months: number analyzed (Participants) | 31 | 29
  2 months | 8.84 (3.45) | 8.90 (5.31)
  4 months: number analyzed (Participants) | 31 | 29
  4 months | 8.52 (4.62) | 7.10 (4.80)
  6 months: number analyzed (Participants) | 30 | 28
  6 months | 8.16 (5.52) | 6.35 (4.49)
  8 months: number analyzed (Participants) | 30 | 28
  8 months | 6.70 (2.90) | 6.33 (3.88)
Statistical Analysis 1: Comparison: Pregnancy Skills Group; We used multilevel generalized mixed modeling under an intent-to-treat approach to compare the outcome measures of EPDS between group 1 (VCI) and Group 2 (AC) at 6 time points during pregnancy and postpartum controlling for screening EPDS score. We powered for the fixed effect of Intervention X Time using RMANOVA with alpha = 0.5, 6 time points, 0.3 for correlation between repeated measures, and a sample size of 192 total participants gives greater than 90% power to detect an effect size of 0.1; Test type: Other — Mean differences at the tested timepoints between VCI and AC. Models were also examined with the covariates of medication use and pregnant/post-partum status; p = 0.612, Mixed Models Analysis; Mean estimates by time = 0.913, 95% CI 2-sided [-1.228 to 3.055], Standard Error of Mean 1.085 — Time was treated as a categorical variable to allow for non-linear change over time. We present group, time, and group*time estimates and their associated SE and CIs below. AC group and baseline timepoint are the reference categories; Overall test of significance for Fixed Effects. Higher EPDS scores signify worsened symptoms of depression. Time uses start of study as reference controlling for screen EPDS. Group VCI (AC reference): F=0.260, p=0.612 Time (Baseline as reference): F=9.021, p<0.001 Group*Time: F=0.537, p=0.748 Estimates for group, time, and group*time interactions Group: Estimate=0.913 (SE=1.085) [CI LB=-1.228, UB=3.055] Time: Post: estimate=-2.766 (0.853) [-4.445, -1.087] 2 months: estimate=-1.517 (0.862) [-3.214, 0.180] 4 months: estimate=-3.186 (0.862) [-4.883, -1.489] 6 months: estimate=-2.781 (0.872) [-4.498, -1.065] 8 months: estimate=-3.103 (0.872) [-4.819, -1.386] Group*Time: Post: estimate=-1.157 (1.214) [-3.547, 1.232] 2 months: estimate=-1.361 (1.210) [-3.742, 1.019] 4 months: estimate= 0.183 (1.209) [-2.196, 2.562] 6 months: estimate=-0.508 (1.223) [-2.914, 1.898] 8 months: estimate=-0.127 (1.220) [-2.529, 2.275]

2. Secondary Outcome: Change in Anxiety Symptoms Over Time
Description: Self-completed: Generalized Anxiety Disorder - 7 Item scale measures symptoms of anxiety. The instrument will measures anxiety symptoms at 6 time points during pregnancy and postpartum. The instrument is on a scale of 0-21, with 0 indicating no symptoms, and 21 indicating the highest severity of symptoms. Scores of < 5 = no anxiety; 5-9 = mild; 10-14 = moderate; > 15 = severe.
Time Frame: Time 1 = pre-intervention; T2 = immediately following week 9 of group intervention classes (post-intervention), T3= 2 months post-intervention; T4= 4 months post-intervention; T5 = 6 months post-intervention; T6 = 8 post-intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | UPLIFT Program | Pregnancy Skills Group
Number analyzed (Participants) | 40 | 41
units on a scale
  Baseline: number analyzed (Participants) | 36 | 33
  Baseline | 6.97 (3.01) | 6.97 (3.01)
  Post: number analyzed (Participants) | 29 | 30
  Post | 5.17 (3.34) | 5.17 (3.34)
  2 months: number analyzed (Participants) | 31 | 29
  2 months | 6.31 (4.04) | 6.31 (4.04)
  4 months: number analyzed (Participants) | 31 | 29
  4 months | 5.45 (3.34) | 5.45 (3.34)
  6 months: number analyzed (Participants) | 30 | 28
  6 months | 4.74 (4.18) | 4.74 (4.18)
  8 months: number analyzed (Participants) | 30 | 28
  8 months | 4.35 (2.68) | 4.35 (2.68)
Statistical Analysis 1: Comparison: Pregnancy Skills Group; We used multilevel generalized mixed modeling under an intent-to-treat approach to compare the outcome measures of GAD-7 between group 1 (VCI) and Group 2 (AC) at 6 time points during pregnancy and postpartum. We powered for the fixed effect of Intervention X Time using RMANOVA with alpha = 0.5, 6 time points, 0.3 for correlation between repeated measures, and a sample size of 192 total participants gives greater than 90% power to detect an effect size of 0.1; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.558, Mixed Models Analysis; Mean estimates by time = 0.0160, 95% CI 2-sided [-1.709 to 1.677], Standard Error of Mean 0.859 — [estimate comment as in outcome 1, analysis 1]; Overall test of significance for Fixed Effects. Higher GAD-7 scores signify worsened symptoms of depression. Group VCI (AC reference): F=0.347, p=0.558 Time (Baseline as reference): F=4.973, p<0.001 Group*Time: F=0.417, p=0.837 Estimates for group, time, and group*time interactions Group: Estimate=-0.0160 (SE=0.859) [CI LB=-1.709, UB=1.677] Time: Post: estimate=-1.780 (0.708) [-3.173, -0.387] 2 months: estimate=-0.615 (0.715) [-2.023, 0.792] 4 months: estimate=-1.416 (0.715) [-2.824, -0.008] 6 months: estimate=-1.625 (0.723) [-3.049, -0.201] 8 months: estimate=-1.542 (0.723) [-2.966, -0.118] Group*Time: Post: estimate=-1.157 (1.214) [-3.547, 1.232] 2 months: estimate=-1.361 (1.210) [-3.742, 1.019] 4 months: estimate= 0.183 (1.209) [-2.196, 2.562] 6 months: estimate=-0.508 (1.223) [-2.914, 1.898] 8 months: estimate=-0.127 (1.220) [-2.529, 2.275]

ADVERSE EVENTS:
Time Frame: Participant data was collected over 10 months from start of intervention.
Description: EPDS scores were monitored for scores over 20. While an EPDS score of >20 indicates a higher risk of depression and anxiety, IRB didn't considered this to be an adverse event given the target population and inclusion criteria. Participants who scored above 20 were referred to a licensed mental health professional for immediate follow-up. During sessions, facilitators also monitored participants' progress and signs they may be considering self-harm.
Arm/Group | UPLIFT Program | Pregnancy Skills Group
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/41
Other Adverse Events (participants affected / at risk) | 0/40 | 0/41

LIMITATIONS AND CAVEATS:
Limitations included low recruitment (largely due to COVID-19), difficulty in identifying participation in either group as the cause of lower EPDS scores 8 months after participation, and difficulty in accounting for factors impacting personal changes that can occur in the 10 months of involvement in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/60/NCT03932760/Prot_SAP_002.pdf
  • Informed Consent Form (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT03932760/ICF_003.pdf